CLINICAL TRIAL: NCT07281781
Title: Treating Anemia in Myelofibrosis With Repurposed Drugs (Nelfinavir) That Restore Iron Delivery to the Bone Marrow
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Angela G. Fleischman, Associate Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6408; UCI 22-118 (Other: UCI CFCCC)
Record Dates: First submitted 2025-12-04; First posted 2025-12-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Myelofibrosis; Myelofibrosis; Anemia
Keywords: Myelofibrosis; Anemia; Nelfinavir
MeSH Terms: conditions — Primary Myelofibrosis; Anemia | interventions — Nelfinavir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nelfinavir (Experimental): Given Orally
  Interventions: Drug: Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir — Taken twice daily

SUMMARY:
This is a phase I/II protocol investigating whether Nelfinavir can improve anemia and lower serum fibrosis biomarkers in Myelofibrosis patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Have a diagnosis of myelofibrosis (MF) according to the 2016 WHO criteria
* Has a hemoglobin ≤ 10gm/dL at screening
* Serum ferritin ≥ 100
* May continue on current MPN treatment, including aspirin, hydroxyurea, interferon-alpha, ruxolitinib, fedratinib, or anagrelide.
* Peripheral blast count <10% during Screening.
* Free of other known active or metastatic malignancies other than localized skin cancer.
* Amenable to blood draws and symptom assessments.
* Agree to the use of contraceptives. Female subjects of childbearing potential and their male partners, or male subjects who have female partners of childbearing potential, should both use an effective contraception method during the study and continue to use contraception for 60 days after the last dose of study drug.

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) questionnaire score of ≥3
* Currently pregnant or planning on being pregnant within the study period.
* Currently taking Momelotinib or Pacritinib (these agents are purported to reduce hepcidin).
* Currently taking any of the contraindicated medications to Nelfinavir listed in section 13.2
* Currently breastfeeding.
* Known uncontrolled active viral or bacterial infection.
* Known HIV+
* Significant impairment of major organ or hematopoietic function defined as

  1. Serum creatinine clearance less than 30 ml/min (eGFR).
  2. Bilirubin more than 1.5 mg/dl except for Gilbert's disease. ALT or AST more than 2X upper normal limit or has radiologic evidence of liver cirrhosis.
  3. Platelets < 50 × 10^9/L without transfusions
  4. ANC < 0.75 × 10^9/L without growth factors
* Known history of allergic reaction to nelfinavir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Hepcidin Levels | 30 days
  Comparison of Hepcidin Levels prior to and after Nelfinavir treatment

SECONDARY OUTCOMES:
Change in Hemoglobin Levels | 30 days
  Comparison of hemoglobin levels to determine whether there is restoration of iron to the bone marrow.
Change in Fibrosis Biomarkers | 30 days
  To evaluate if nelfinavir lowers fibrosis biomarkers in serum.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Flesichman, MD, PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States